CLINICAL TRIAL: NCT04062006
Title: Low-dose Interleukin-2 Treatment on Polymyalgia Rheumatica
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-PHB089-03
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interleukin-2 (Experimental): low dose interleukin-2 injected subcutaneously, at a dose of 1 x 10~6 IU/m2 five days per week for 4 weeks (day1-5, 8-12, 15-19, 22-26) and then once a week for 8 weeks (day33, 40, 47, 54, 61, 68, 75, 82).
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — low dose interleukin-2 injected subcutaneously, at a dose of 1 x 10~6 IU/m2 five days per week for 4 weeks (day1-5, 8-12, 15-19, 22-26) and then once a week for 8 weeks (day33, 40, 47, 54, 61, 68, 75, 82).
  Other Names: Recombinant Human Interleukin-2

SUMMARY:
This study aims to explore the clinical and immunological efficacy of low-dose Interleukin-2 (IL-2) on polymyalgia rheumatica.

DETAILED DESCRIPTION:
The investigators designed a single center, open-label, prospective study that routinely administered low-dose IL-2 therapy to monitor the improvement of clinical and laboratory parameters to explore its efficacy and to observe changes in immune cell subsets and cytokines. One million units of Recombinant Human Interleukin-2 (rhIL-2) was administered subcutaneously five days every week for 4 weeks and then once a week for 8 weeks. All patients were followed up for 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥50 years at screening visits
2. Diagnostics meet the 1986 Nancy recommendations
3. Apply glucocorticoids (≤10 mg/d prednisone or equivalent doses of other hormones), DMARDs (eg methotrexate, hydroxychloroquine, azathioprine, morphine, Ester, leflunomide, cyclosporine, etc.) must be stable for 4 weeks and do not increase hormone doses or other immunosuppressive agents throughout the study. If the enrolled doctor plans to stop using the current immunosuppressant or glucocorticoid, the elution period needs to be followed before enrollment. Each drug needs to meet the following elution period

   * Glucocorticoid-2 weeks
   * Immunosuppressants (including methotrexate, azathioprine, cyclosporine, tacrolimus, leflunomide, mycophenolate mofetil) - 4 weeks
   * Intravenous immunogloblin (IVIg) or cyclophosphamide - 2 months
   * Rituximab - 6 months
   * Other biological agents (infliximab, adalimumab, etanercept, anakinra, etc.) -12 weeks
4. The patient must be informed in writing of the consent to participate in the trial and the patient is expected to be able to comply with the requirements of the study follow-up plan and other protocols.
5. Excluding Horton syndrome
6. The amount of non-steroidal dose was stable 4 weeks before enrollment

Exclusion Criteria:

Any subject meeting any of the following criteria should be excluded:

1. Use rituximab or other monoclonal antibodies within 6 months.
2. Received high doses of glucocorticoid (>10 mg/d) within 1 month.
3. Serious complications: including heart failure (≥ New York Heart Association (NYHA) class III), renal insufficiency (creatinine clearance ≤ 30 ml/min), liver dysfunction (serum Alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than three times the upper limit of normal, or total bilirubin greater than Normal upper limit)
4. Other serious, progressive or uncontrollable hematology, gastrointestinal, endocrine, pulmonary, cardiac, neurological or brain disorders (including demyelinating diseases such as multiple sclerosis).
5. Known allergies, hyperreactivity or intolerance of IL-2 or its excipients.
6. Have a serious infection needing hospitalization (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, EB virus, tuberculosis infection), or use intravenous antibiotics to treat infection in 2 months before the enrollment.
7. Chest imaging showed abnormalities in malignant tumors or current active infections (including tuberculosis) within 3 months prior to the first use of the study drug.
8. Infection with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, it is recommended to consult a doctor who has expertise in treating HIV or hepatitis C virus infection.
9. Any known history of malignancy in the past 5 years (except for non-melanoma skin cancer, non-melanoma skin cancer or cervical tumor without recurrence within 3 months after surgical cure prior to the first study preparation).
10. Uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past 3 years, may hinder the successful completion of the study.
11. Accept or expect to receive any live virus or bacterial vaccination within 3 months prior to the first injection of the study agent, during the study period, or within 4 months after the last injection of the study agent. Bacillus Calmette-Guerin (BCG) vaccine was inoculated within 12 months after screening.
12. Pregnant, lactating women (WCBP) are reluctant to use medically approved contraceptives during treatment and 12 months after treatment.
13. Men whose partners have fertility potential but are reluctant to use appropriate medically-accepted contraceptives during treatment and 12 months after the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08-31 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Foxp3+Treg cells: change in percentage of total lymphocytes | week 12
  Treg refers to regulatory T cells

SECONDARY OUTCOMES:
Physician's Global Disease Activity VAS | week12 and 24
  Physician's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the polymyalgia rheumatica).
Patient's Global Disease Activity VAS | week12 and 24
  Patient's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the polymyalgia rheumatica).
Safety and tolerability of interleukin-2 as assessed by incidence of adverse events reported and observed | up to 24 weeks
  The investigators will report frequency of adverse events
Patient reported outcome 36-item Short Form Health Survey (SF-36) | wee12 and 24
  Clinical studies 36-item Medical Outcomes Study Short-Form General Health Survey An instrument used to assess multidimensional health-related quality of life (QOL), which measures 8 health related parameters: physical function, social function, physical role, emotional role, mental health, energy, pain, general health perceptions; each parameter is scored from 0 to 100 Managed care 36-Item Short-Form Functional and Perceived Health Status Survey A questionnaire which measures health status; the SF-36 also includes a list of 18 self-reported chronic conditions
Proportion of patients with Low disease activity (PMR-AS<10) with steroid independence (GCs ≤5 mg absolute value) or decrease ≥ 10 mg | from week 0 to week 12 and 24
  PMR-AS was developed from the following components: measure of C-reactive protein (CRP), measure of Erythrocyte Sedimentation Rate (ESR), assessment of early morning stiffness, assessment of the patient's elevation on upper limbs, patient's assessment of pain, and physician's global assessment of disease activity.
Cumulative dosages of glucocorticoids (GCs) | week 12 and 24
  dosages of GCs
The proportion of patients with PMR-activity score (AS) < 1.5; 10; 17 | week 12 and 24
  PMR-AS was developed from the following components: measure of C-reactive protein (CRP), measure of Erythrocyte Sedimentation Rate (ESR), assessment of early morning stiffness, assessment of the patient's elevation on upper limbs, patient's assessment of pain, and physician's global assessment of disease activity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kermani TA, Warrington KJ. Advances and challenges in the diagnosis and treatment of polymyalgia rheumatica. Ther Adv Musculoskelet Dis. 2014 Feb;6(1):8-19. doi: 10.1177/1759720X13512450. PMID 24489611
- [Result] Brooks RC, McGee SR. Diagnostic dilemmas in polymyalgia rheumatica. Arch Intern Med. 1997 Jan 27;157(2):162-8. PMID 9009973
- [Result] Bird HA, Esselinckx W, Dixon AS, Mowat AG, Wood PH. An evaluation of criteria for polymyalgia rheumatica. Ann Rheum Dis. 1979 Oct;38(5):434-9. doi: 10.1136/ard.38.5.434. PMID 518143